CLINICAL TRIAL: NCT06942299
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Pharmacokinetics, Safety, and Efficacy of Multiple Doses AK0529 in Adult Hospitalized Subjects With Respiratory Syncytial Virus Infection
Brief Title: A Study of AK0529 in Adults Patients Hospitalized With RSV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK0529-2005
Record Dates: First submitted 2023-03-24; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Adult patient with RSV infection; High-risk disease; AK0529
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — ziresovir

STUDY DESIGN:
Intervention Model Description: This clinical study is a randomized placebo controlled parallel multi-center phase II trial.
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active drug: AK0529 fasting (Experimental): The participants will receive AK0529 twice daily for 5 days from D1 to D5.
  Interventions: Drug: AK0529
- Active drug: AK0529 with meal (Experimental): The participants will receive AK0529 twice daily for 5 days from D1 to D5.
  Interventions: Drug: AK0529
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK0529 — Active Substance: AK0529, Pharmaceutical Form: Enteric pellets, Route of Administration: Oral, fasting
  Arms: Active drug: AK0529 fasting
Drug: AK0529 — Active Substance: AK0529, Pharmaceutical Form: Enteric pellets, Route of Administration: Oral with meal
  Arms: Active drug: AK0529 with meal
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Enteric pellets, Route of Administration: Oral with meal or fasting
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, phase II study to be conducted in adults hospitalized with RSV infection in China. The main objectives of this study are to investigate the safety, pharmacokinetics and efficacy of AK0529 in adult RSV patients.

ELIGIBILITY:
Main Inclusion criteria:

1. . Male or female patients of any ethnicity with an age of 18-85 years.
2. . Diagnosis of RSV infection by any virological means within 36 hours preceding initial dosing.
3. . At least one of the following high-risk diseases or states for RSV infection

   1. Asthma or chronic lung disease (such as COPD or cystic fibrosis),
   2. immunocompromised,
   3. Heart disease (such as congenital heart disease, congestive, heart failure, or coronary artery disease), except high blood, pressure without heart-related symptoms,
   4. Chronic kidney disease,
   5. Age ≥65 years old.
4. . With at least 1 new onset respiratory infection symptom or exacerbation of existing respiratory symptoms (respiratory symptoms include: sore throat, nasal congestion, runny nose, sneezing, coughing, wheezing, sputum production, shortness of breath), and any individual score is 2 or moderate.
5. . Onset of RSV infection symptoms should be ≤ 7 days.

Main Exclusion criteria:

1. . 3 days for drugs with potential antiviral effects on RSV such as ordinary interferon, 8 days for long-acting interferon, and 35 days for ribavirin for 5 half-lives before expected administration.
2. . Prohibited medicine are being used or planned to be used during the study treatment periods.
3. . Severe gastrointestinal diseases that affect the absorption of study drugs (such as vomiting, malabsorption syndrome, short bowel syndrome due to necrotizing enterocolitis, etc.).
4. . Received or planned to have bone marrow transplantation, stem cell transplantation or solid organ transplantation within 1 year.
5. . Patients with malignant tumors who had surgery within recent 6 months and/or requiring radiotherapy, chemotherapy and biological immunotherapy.
6. . Patients with autoimmune diseases who are in the induction treatment.
7. . HIV infection, CD4 count< 350 cells/mm3 with opportunistic infection and need treatment.
8. . Other patients who are judged by the investigator to be unsuitable for participating in the study, such as acute/chronic heart, lung, liver, kidney, rheumatic immunity, psychiatric, blood and other diseases in the unstable period.
9. . History of drug abuse within 12 months prior to screening.
10. . Allergy to the investigational drug or its component.
11. . Female patients with positive pregnancy test or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AE and SAE of subjects during the study period | Baseline up to 28 days
  An Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect, or another important medical event.

SECONDARY OUTCOMES:
Change from baseline in clinical improvement score of subjects at each visit after treatment by clinical improvement scale | Baseline up to 28 days
  Clinical improvement scale is mainly used to evaluate the overall severity level of the subject's disease with the highest score of 8 indicating death. A score of 6-7 represents severe hospitalization: a score of 6 requires mechanical ventilation, and a score of 7 requires not only mechanical ventilation but also angiogenic treatment, kidney dialysis, or artificial membrane lung. A score of 3-5 represents mild hospitalization: a score of 3 does not require oxygen therapy, a score of 4 requires a mask or nasal catheter, and a score of 5 requires noninvasive positive pressure ventilation or high-flow oxygen therapy. A score of 1-2 represents outpatient treatment: 1 is independent and 2 is in need of care (daily activities have an impact). A score of 0 means no treatment is required and there is no clinical or virological evidence of infection.
Change from baseline in RiiQ symptoms of subjects at each visit after treatment measured by RiiQ questionnaire | Baseline up to 28 days
  RiiQ questionnaire is mainly used to assess RSV symptoms in patients, including upper respiratory tract infection symptoms (sore throat and nasal congestion), symptoms of lower respiratory tract infection (cough, wheezing, sputum, shortness of breath), and system symptoms (fever, headache, neck pain, fatigue, lack of appetite, interrupted sleep, body aches). The questionnaire is divided into four grading categories of severity including none (0), mild (1), moderate (2) and severe (3).
Changes from baseline in the total score of RSV Symptom of subjects at each visit after treatment using RSV Symptom Score Composite Scale | Baseline up to 28 days
  RSV Symptom Score Composite Scale is used to assess patients with RSV symptoms, including runny nose, stuffy nose, sneezing, sore throat, earache, cough, shortness of breath, headache, fatigue, myalgia and/or joint pain. The score is divided into 4 grades according to the severity of symptoms. 0 indicates no symptoms, 1 indicates occasional symptoms, 2 indicates that symptoms sometimes worsen significantly but do not affect daily activities, and 3 indicates that symptoms are always serious and cannot engage in daily activities. The total score is 30 points.
Changes from baseline in the RSV VL (viral load) of subjects at each visit after treatment | Baseline up to 28 days
  The RSV VL of subjects' nasopharyngeal samples is measured as Log10 copies/mL by quantitative reverse transcription polymerase chain reaction (qRT-PCR).
Area under the curve (AUCE, last) of RSV Viral Load from baseline to the last measurement | Baseline up to 28 days
  The RSV VL is measured as Log10 copies/mL by qRT-PCR assay in the nasopharyngeal specimens.
Number of subjects with RSV VL values below the lower limit of quantitation (LLOQ) at each visit after treatment | Baseline up to 28 days
  The RSV VL is measured as Log10 copies/mL by qRT-PCR assay in the nasopharyngeal specimens.
Number of participants who dropped out of the study due to AE | Baseline up to 28 days
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Number of participants with laboratory examination abnormalities | Baseline up to 28 days
  Following parameters were analyzed for laboratory examination: hemoglobin (Hb), hematocrit, platelet count, red blood cell (RBC) count, white blood cell (WBC) count, mean corpuscular volume (MCV) and absolute white blood cell line (neutrophils, eosinophils, lymphocytes, monocytes, basophils); Hepatobiliary biochemistry: total and direct bilirubin, total protein, albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP); Renal Function Tests: creatinine kinase, uric acid ; Electrolytes: Sodium, Potassium; Glucose; Coagulation function (subjects with only a history of liver disease should be tested): international normalized ratio (INR), activated partial thromboplastin time, prothrombin time, thrombin time, and fibrinogen; Urine analysis: urine protein, ketone bodies, urine red blood cells, urine white blood cells, and urine glucose; Blood or urine pregnancy test for all female subjects.
Number of participants with vital sign abnormalities | Baseline up to 28 days
  Number of participants with vital sign (systolic and diastolic blood pressure, pulse rate, respiratory rate, temperature and oxygen saturation) abnormalities were reported.
Number of participants with physical examination abnormalities | Baseline up to 28 days
  A comprehensive physical examination includes at least cardiovascular, respiratory, gastrointestinal, and nervous system assessments; a simple physical examination includes at least skin, lung, cardiovascular system and abdominal (liver and spleen) assessments.
Number of participants with ECG abnormalities | Baseline up to 28 days
  Electrocardiograms were measured during the screening period, at 4 (±1) hours after the first dose on day 2, at 4 (±1) hours and 12 (±1) hours (before the second dose) after the first dose on day 4, and once on day 6 and day 14 during the follow-up period; 9-or 12-lead ECG results are recorded using an ECG instrument which automatically calculates heart rate and measures PR, QRS, QT and QTc intervals.
Peak Plasma Concentration (Cmax) | Day 1, Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.
Time to Maximum Plasma Concentration (Tmax) | Day 1，Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.
Terminal Elimination Half-life (t½) | Day 1，Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.
Apparent Clearance (CL/F) | Day 1，Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.
Apparent Volume of Distribution (V[z]/F) | Day 1，Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.
Area Under the Plasma Concentration-Time Curve From Time 0 to 12 (AUC[0-12]) | Day 1，Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.
Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC[0-∞]) | Day 1，Day 5
  Whole blood of subjects (2 mL per time point) was collected for the concentration determination of the AK0529 and its metabolites at various time points on day 1 and day 5, and the PK parameter is calculated using the above-mentioned plasma concentration data.

CONTACTS AND LOCATIONS:
Locations (42):
- China (42):
  - The Second Perople's Hospital of Hefei, Hefei, Anhui
  - Huangshan City People's Hospital, Huangshan City, Anhui
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Gansu People's Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Longgang Central Hospital of Shenzhen, Shenzhen, Guangdong
  - Shunde Hospital of Southern Medical University, Shunde, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - The Second Nanning People's Hospital, Nanning, Guangxi
  - Guizhou People's Hospital, Guiyang, Guizhou
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Affiliated Fourth Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Heilongjiang University of Traditional Chinese Medicine, Harbin, Heilongjiang
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Wuhan Fourth Hospital, Wuhan, Hubei
  - Xiangyang Center Hospital, Xiangyang, Hubei
  - Yueyang Central Hospital, Yueyang, Hunan
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - Jiangsu Provincial Hospital of Chinese Medicine, Nanjing, Jiangsu
  - The First Affilited Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Clinical College / Liaoning Hospital of TCM, Shenyang, Liaoning
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Neimenggu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang NO.2 People's Hospital, Weifang, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Yueyang Hospital Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Sencond Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - Chengdu Seventh People's Hospital, Chengdu, Sichuan
  - The First Hospital of Kunming, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No